CLINICAL TRIAL: NCT00120666
Title: Interhemispheric Plasticity in Humans
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050188; 05-N-0188
Record Dates: First submitted 2005-07-16; First posted 2005-07-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-06-25

CONDITIONS: Healthy
Keywords: Exercise; Stimulation; Nerve; Electrical; Muscle; Healthy Volunteer; HV
MeSH Terms: conditions — Motor Activity

SUMMARY:
This study will determine how the brain controls movements by sending messages to the spinal cord and muscles. Researchers want to know if strengthening a hand muscle will increase the strength of the same muscle in the other hand, and if these changes happen in the brain or spine, or both. Plasticity in this study refers to the capacity for continuous changes of the neural pathways in the brain and nervous system. Researchers have seen cases in which using a muscle extensively (force production) in one muscle group has increased the strength of the same muscle group on the opposite side of the body (force transfer). This situation happens without the unused muscle becoming larger-suggesting that the practice causes changes in some parts of the brain or spine. It is vital for scientists to know how this effect works, so that they can create new rehabilitation methods for people who cannot move or who have difficulty moving one side of their body.

Patients ages 18 to 60 who are in good health and who do not have a history of major conditions affecting the bones, joints or nervous system may be eligible for this study. Patients will undergo a medical examination. There will be 1 or 2 testing sessions, 20 training sessions, and 1 or 2 final testing sessions, with patients being asked to come to the laboratory for as few as 4 times (about 10 hours total) or for up to 25 visits (about 20 hours total). The investigator will indicate which of six different groups that a patient is selected for.

During testing sessions, the strength of the pointer and little fingers in each hand will be determined through the use of very brief electrical pulses. There also will be transcranial magnetic stimulation (TMS) and 1 Hz TMS. The researchers will place one or two wire coils on the patient's scalp and make marks on the scalp which will be removed at the end of the session. During the TMS, a brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. Patients will hear a click sound and feel a snapping sensation on the skin. They may also feel and see small twitches in the hand muscles, and the fingers or wrist may move. There will be a total of about 300 magnetic stimuli, at a rate of 10 pulses per minute. Patients will also have an electromyogram (EMG), a procedure recording electrical activity in the muscles that are activated by electrical or magnetic stimulation. Metal electrodes will be attached to the skin over the muscle. During the EMG, patients will be asked to tense certain muscles slightly. Depending on the group a patient is assigned to, he or she may be asked to use the right index finger by using voluntary muscle movement, electrical stimulation, his or her imagination, electrical stimulation of a different hand muscle, or voluntary movements immediately followed by repetitive TMS.

Regardless of group assignment, there will be five blocks of 10 repetitions of finger exercise per session, 200 per week, and 1,000 throughout the whole study. During the study sessions, patients will be able to talk and move around. They can take a break and leave the room if needed. In most cases, the session will take less than 2 hours. There also will be a control group whose members will not be training their fingers but who will participate only in the testing sessions. TMS is a safe procedure; however, strong contractions of scalp muscles have been known to cause headaches. Also, because of the distracting noise of the TMS, patients will be fitted with earplugs to wear during the procedure.

Compensation for research-related discomfort and inconvenience will be made to participants, with a maximum of $500 to $600, depending on assignment to groups. This study will not have a direct benefit for participants. However, researchers hope to gain information that will help them better understand how the two sides of the brain control movement and how they affect each other regarding movement control.

DETAILED DESCRIPTION:
Strength training of a limb muscle on one side of the body produces functionally and clinically meaningful increases in motor output of the same muscle on the opposite side of the body. Such adaptations occur without muscle hypertrophy, implying a role for the ipsilateral motor cortex and the spinal cord in force transfer. The goal of this project is to determine the interhemispheric and spinal mechanisms of force transfer in healthy young adults. We hypothesize that the effects of unilateral practice on interhemispheric inhibition (IHI) and on the excitability of the contralateral corticospinal projections are linked, and these effects are graded according to the nature of muscle activation. In a series of experiments on healthy adults age 18 to 60, we will characterize the motor cortical inhibitory and excitatory mechanisms of interhemispheric practice-induced transfer of muscle force.

We will use a longitudinal design that will include three exercise groups. In 20 sessions over 4 weeks, subjects will strengthen their first dorsal interosseus (FDI) muscle of the dominant hand either with voluntary, electrically stimulated, or imagined contractions. The design also includes three control groups, a sham-stimulated group, a repetitive transcranial magnetic stimulation (1HzTMS) group, and a no-intervention group. Before and after the training programs, we will determine the changes in the outcome measures, including voluntary and electrical stimulation evoked force of the trained and the untrained FDI. Measures of excitability of the involved and uninvolved motor cortex, assessed with TMS, and measures of spinal cord excitability, assessed with peripheral nerve stimulation, are the additional outcome measures. The results of these studies will substantially increase our understanding of central nervous system (CNS) control of voluntary movement in health and disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Male and female volunteers ages 18-60 years old will qualify for this study. The subject population will be equitable and we will strive to enroll volunteers from all ethnic backgrounds.

EXCLUSION CRITERIA:

1. orthopedic impairments of the upper extremities
2. neurological impairments, including current or past peripheral or central nervous system dysfunction
3. being on drugs that may lower the seizure threshold
4. having a pacemaker, an implanted medication pump, a metal plate in the skull, metal objects in the eye or skull (for example after brain surgery or shrapnel wounds)
5. consumption of more than moderate amounts of alcohol or caffeine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108
Dates: Start 2005-07-08; Study Completion 2007-06-25

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] ASANUMA H, OKUDA O. Effects of transcallosal volleys on pyramidal tract cell activity of cat. J Neurophysiol. 1962 Mar;25:198-208. doi: 10.1152/jn.1962.25.2.198. No abstract available. PMID 13862744